CLINICAL TRIAL: NCT00693199
Title: Effect of Amlodipine Monotherapy or Combined With Terazosin on Lower Urinary Tract Symptoms and Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anhui Medical University (Other)
Collaborators: The University of Science and Technology of China (Other); Peking University First Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BMI-AT-02
Record Dates: First submitted 2008-06-05; First posted 2008-06-06 (Estimated); Last update posted 2008-08-08 (Estimated); Status verified 2008-06

CONDITIONS: Lower Urinary Tract Symptoms; Hypertension
Keywords: Amlodipine; Terazosin; Lower Urinary Tract Symptoms (LUTS); Essential hypertension; International Prostate Symptom Score (IPSS); Quality Of Life (QOL)
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Hypertension; Essential Hypertension | interventions — Amlodipine; Terazosin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: amlodipine
- 2 (Active Comparator)
  Interventions: Drug: terazosin
- 3 (Experimental)
  Interventions: Drug: amlodipine plus terazosin

INTERVENTIONS:
Drug: amlodipine — amlodipine 5mg once daily for 28 days
  Arms: 1
Drug: terazosin — terazosin 2 mg once daily for 28 days
  Arms: 2
Drug: amlodipine plus terazosin — amlodipine 5 mg plus terazosin 2 mg once daily for 28days
  Arms: 3

SUMMARY:
The aim of this study was to investigate the efficacy and safety of low dose amlodipine alone, or combined with low dose terazosin in male patients with both lower urinary tract symptoms and hypertension.

ELIGIBILITY:
Inclusion Criteria:

1. Men 50 years or older
2. with LUTS [defined as International Prostate Symptom Score (IPSS) >= 10].
3. Stage 1 or 2 essential hypertension (SBP >= 140 mm Hg and < 180 mm Hg and/or DBP >= 90 mm Hg and < 110 mm Hg)

Exclusion Criteria:

1. A history of postural hypotension
2. Secondary hypertension
3. Prostate cancer
4. Prostate surgery or other intervention
5. Use of any agents to influence the LUTS symptoms in the last 4 weeks
6. Other severe diseases

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2006-07; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
The primary efficacy outcomes were reductions in blood pressure and International Prostate Symptoms Score (IPSS) and sub-scores. | 28th day after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ping Liu, PhD, Study Director — Biomedical Institute of Anhui Medical University
Locations (1):
- Biomedicine Inistitute of Anhui Medical University, Hefei, Anhui, China

REFERENCES:
- [Derived] Liu H, Liu P, Mao G, Chen G, Wang B, Qin X, Na Y, Liu Z, Wang X, Xu X. Efficacy of combined amlodipine/terazosin therapy in male hypertensive patients with lower urinary tract symptoms: a randomized, double-blind clinical trial. Urology. 2009 Jul;74(1):130-6. doi: 10.1016/j.urology.2008.11.051. Epub 2009 Apr 15. PMID 19371934